CLINICAL TRIAL: NCT01345513
Title: Feasibility Clinical Study of Targeted and Genome-Wide Sequencing
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: TGWS-001
Record Dates: First submitted 2011-04-21; First posted 2011-05-02 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Solid Tumors
Keywords: Genomic Analysis; Sequencing; Genetic; Biopsy; Solid tumors
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Archival tumor tissue, fresh tumor biopsy, blood sample, pleural effusion (if available)or ascites (if available)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Solid Tumor Cancer
  Interventions: Other: Sample Collection for Genome-Wide Sequencing

INTERVENTIONS:
Other: Sample Collection for Genome-Wide Sequencing — Collection of archival tumor tissue, fresh tumor biopsy, blood sample, and pleural effusion (if available)or ascites (if available)

SUMMARY:
This research is being done to find out what types of gene mutations are present in people with cancer. This study is designed to help researchers and doctors understand more about cancer. With this information, doctors may have a better idea as to which cancer treatments are most appropriate for certain patients. The information will also help researchers find out the how to identify genes in cancers from biopsies and blood samples and how to use this information to help doctors and patients make treatment decisions.

DETAILED DESCRIPTION:
This is a prospective cohort study with the goal of obtaining fresh tumor biopsies and one blood sample from patients with a confirmed histological or cytological diagnosis of cancer, who are potential candidates for a phase I or II clinical trial at their local institution. DNA from fresh tumor biopsies and from mononuclear blood cells will be subjected to targeted and genome-wide sequencing to enable molecular characterization of tumors. Application of genomic information by investigators will be captured. Archived tumor samples will be requested from all patients. For patients with malignant ascites or pleural effusions, fluid and tumor samples will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Histological or cytological proof of solid tumour cancer.
* At least one biopsiable lesion deemed medically accessible and safe to biopsy.
* Candidate for one or more phase I or II clinical trials in the local institution or in another Ontario institution, at the time of study enrollment or at a later time point.
* Fulfills local institution's laboratory parameters for tumor biopsy.
* Willingness and ability of patient to provide signed voluntary informed consent.

Exclusion Criteria:

* Any condition that could interfere with their ability to provide informed consent such as dementia or severe cognitive impairment.
* Any contraindication to undergoing a biopsy procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Princess Margaret Hospital or other Ontario Institution
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2013-03-25 (Actual); Study Completion 2019-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Solid Tumor Cancer
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Of the 56 participants approached, 50 agreed and consented to the study, and 49 had successful biopsies.
Arm/Group | Solid Tumor Cancer
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 57 [44 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Time Since Metastatic Diagnosis (Months) [Median (Full Range); unit: months] | 17.2 [1.2 to 81.8]
Number of Prior Treatment Regimens [Median (Full Range); unit: prior treatment regimens] | 3 [0 to 8]
Primary Tumour Type [Count of Participants; unit: Participants]
  Colorectal | 9
  Breast | 8
  Ovarian | 8
  NSCLC | 5
  Prostate | 3
  Anal | 2
  Mesothelioma | 2
  Head & Neck | 2
  Other | 11

OUTCOME MEASURES:

1. Primary Outcome: Time From Patient Recruitment to Final Results ≤ 21 Days in ≥ 90% of Patients
Description: Average and range of time (in calendar days) that occurred between study participants providing informed consent to the reporting of genomic results to the physician.
Time Frame: All patients will be followed for up to 2 years from study enrolment, or death, or whichever event occurs first.
Measure: Mean (Full Range); unit: calendar days
Arm/Group | Solid Tumor Cancer
Number analyzed (Participants) | 49
calendar days | 21 [7 to 63]

2. Secondary Outcome: Number of Participants With Actionable Genomic Results
Description: Number of participants with actionable genomic results (defined as having the potential to impact on management recommendations based on diagnostic, prognostic and/or predictive implications), expressed as a percentage of the total number of study participants.
Time Frame: All patients will be followed for up to 2 years from study enrolment, or death, or whichever event occurs first.
Measure: Count of Participants; unit: Participants
Arm/Group | Solid Tumor Cancer
Number analyzed (Participants) | 49
Participants | 16

3. Secondary Outcome: Number of Participants With Adverse Events Due to Tumor Biopsies on Study
Description: Number of participants with any adverse events possibly, probably or definitely related to tumor biopsies on study; Grading by CTCAE version 4 of adverse events.
Time Frame: All patients will be followed for up to 2 years from study enrolment, or death, or whichever event occurs first.
Population: Of the 49 patients analyzed, 8 experienced adverse events related to tumour biopsies during the study. Minor events included bruising, bleeding and minor infections. Serious events included pneumothorax and cellulitis.
Measure: Count of Participants; unit: Participants
Arm/Group | Solid Tumor Cancer
Number analyzed (Participants) | 8
Participants
  Minor (as per CTCAE) | 6
  Serious (as per CTCAE) | 2

4. Secondary Outcome: Patient and Physician Experience
Description: Qualitative and quantitative responses on questionnaires and personal interviews regarding patient and physician experience of this research process and their understanding of genomic analysis including perceptions of benefit versus disadvantages, impact on clinical care and decision making
Time Frame: All patients will be followed for up to 2 years from study enrolment, or death, or whichever event occurs first.
Population: Data were not collected.
Arm/Group | Solid Tumor Cancer
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Solid Tumor Cancer
Serious Adverse Events (participants affected / at risk) | 2/49
Other Adverse Events (participants affected / at risk) | 6/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solid Tumor Cancer (N=49)
Grade 2 Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Grade 3 Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solid Tumor Cancer (N=49)
Grade 1 Bruising (Skin and subcutaneous tissue disorders) | 6 (6)
Grade 1 Bleeding (Skin and subcutaneous tissue disorders) | 6 (6)
Grade 2 Wound Infection (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes